CLINICAL TRIAL: NCT01087099
Title: A Multinational Trial of the Efficacy of Albendazole Against Soil-transmitted Nematode Infections in Children
Acronym: WORMCON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: World Health Organization (Other); George Washington University (Other); Commonwealth Scientific and Industrial Research Organisation, Division of Livestock Industries, Brisbane, Australia (Unknown); University of Nottingham (Other); Queensland Institute of Medical Research (Other)
Responsible Party: Jozef Vercruysse, University Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008/322
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-07

CONDITIONS: Infections With Soil-Transmitted Helminths (STH)
MeSH Terms: interventions — Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Albendazole (Experimental): Treatment with albendazole
  Interventions: Drug: Albendazole

INTERVENTIONS:
Drug: Albendazole — Treatment with albendazole

SUMMARY:
The three major Soil-Transmitted Helminths (STH), Ascaris lumbricoides, Necator americanus/Ancylostoma duodenal and Trichuris trichiura are among the most prevalent parasites worldwide. The objective of this multicentre international study is to define the efficacy of a single 400 milligram dose of albendazole (ALB) against these three STHs using a standardised protocol. The trial will be undertaken among school age children in seven countries - Brazil, Cameroon, Cambodia, Ethiopia, India, Tanzania (Zanzibar) and Vietnam - each with a different epidemiologic pattern of infection. A trial of this nature is urgently required because in spite of the wide usage of albendazole over the last 3 decades, there is still no key publication reporting the efficacy of the anthelmintic accurately, and to modern conventional standards, that can act as a central reference for the baseline efficacy. The latter is critically important because albendazole is now being used even more widely, as large scale mass treatment campaigns are being implemented in Africa and elsewhere, with the intention of reducing morbidity in children. Such large scale usage of a drug risks resistance developing, but resistance cannot be detected unless benchmark values for baseline efficacy are widely known.

ELIGIBILITY:
Inclusion Criteria:

* Children should be infected with a minimum of 150 eggs/gram of any of the three species of STH (i.e. Ascaris or hookworms or Trichuris).

Exclusion Criteria:

* Not willing to participate
* Unable to give samples for follow up
* Severe intercurrent medical condition
* Diarrhoea at first sampling

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1750 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of albendazole | 14 to 30 days after treatment
  To determine the efficacy of albendazole, and this will be assessed by the reduction in parasite faecal egg counts between the pre- and post-intervention surveys. The latter will be conducted 14-30 days after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Vercruysse, Principal Investigator — University Ghent
Locations (7):
- Instituto René Rachou, Fundação Oswaldo Cruz, Minas Gerais, Brazil
- Institut Pasteur in Cambodia, Clinical Pathology Unit, Phnom Penh, Cambodia
- Centre for Schistosomiasis and Parasitology, Faculty of Sciences, University of Yaoundé I, Yaoundé, Cameroon
- Department of Medical Laboratory Sciences and Pathology , College of Public Health and Medical Sciences, Jimma University, Jimma, Ethiopia
- Department of Gastrointestinal Sciences, Christian Medical College, Vellore, India
- Public Health Laboratory, Zanzibar, Tanzania
- National Institute for Malariology, Parasitology and Entomology, Hanoi, Vietnam

REFERENCES:
- [Derived] Levecke B, Montresor A, Albonico M, Ame SM, Behnke JM, Bethony JM, Noumedem CD, Engels D, Guillard B, Kotze AC, Krolewiecki AJ, McCarthy JS, Mekonnen Z, Periago MV, Sopheak H, Tchuem-Tchuente LA, Duong TT, Huong NT, Zeynudin A, Vercruysse J. Assessment of anthelmintic efficacy of mebendazole in school children in six countries where soil-transmitted helminths are endemic. PLoS Negl Trop Dis. 2014 Oct 9;8(10):e3204. doi: 10.1371/journal.pntd.0003204. eCollection 2014 Oct. PMID 25299391
- [Derived] Levecke B, Mekonnen Z, Albonico M, Vercruysse J. The impact of baseline faecal egg counts on the efficacy of single-dose albendazole against Trichuris trichiura. Trans R Soc Trop Med Hyg. 2012 Feb;106(2):128-30. doi: 10.1016/j.trstmh.2011.09.007. Epub 2011 Dec 19. PMID 22189084
- [Derived] Vercruysse J, Behnke JM, Albonico M, Ame SM, Angebault C, Bethony JM, Engels D, Guillard B, Nguyen TV, Kang G, Kattula D, Kotze AC, McCarthy JS, Mekonnen Z, Montresor A, Periago MV, Sumo L, Tchuente LA, Dang TC, Zeynudin A, Levecke B. Assessment of the anthelmintic efficacy of albendazole in school children in seven countries where soil-transmitted helminths are endemic. PLoS Negl Trop Dis. 2011 Mar 29;5(3):e948. doi: 10.1371/journal.pntd.0000948. PMID 21468309